CLINICAL TRIAL: NCT00861666
Title: Forgiveness-Based Writing to Prevent Posttraumatic Stress Disorder in OEF/OIF Veterans
Brief Title: Forgiveness-Based Writing to Prevent Post-Traumatic Stress Disorder (PTSD) in Operation Enduring Freedom/Operation Iraqi Freedom (OEF/OIF) Veterans
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: South Central VA Mental Illness Research, Education & Clinical Center (U.S. Federal Agency)
Responsible Party: Catherine Romero Barber, MIRECC affiliate
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H-23892
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Last update posted 2009-06-03 (Estimated); Status verified 2009-06

CONDITIONS: Stress Disorders, Traumatic; Anxiety Disorders; PTSD
Keywords: Forgiveness; Writing; PTSD; OEF; OIF; Veterans
MeSH Terms: conditions — Stress Disorders, Traumatic; Anxiety Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Forgiveness-based Writing (Other)
  Interventions: Behavioral: Forgiveness-Based Writing

INTERVENTIONS:
Behavioral: Forgiveness-Based Writing — Participants will be asked to complete self-report measures during the initial session, will be given writing instructions and will complete the first writing task on-site. The first writing task will focus on describing an offense in which someone hurt or angered the participant, and about which the participant is still hurt and angry.
  Eleven additional writing tasks will be completed at home, three per week for a month. Writing assignments will include topics such as describing thoughts and feelings about the offense, identifying possible motives or mitigating circumstances, identifying benefits of the offense itself, identifying times when one has offended others and how one felt afterwards, identifying benefits of letting go of the offense, and writing a letter to the offender.
  Participants will return each written assignment to the study staff. All participants will be tracked closely by the study coordinator and receive a reminder phone call on the day of each writing task.

SUMMARY:
The purpose of this study is to evaluate a forgiveness-based writing intervention in an open trial with 20 Operation Enduring Freedom/Operation Iraqi Freedom (OEF/OIF) veterans who have recently experienced combat-related trauma to:

1. Determine the feasibility of delivering the intervention.
2. Evaluate the acceptability of the intervention.
3. Collect preliminary outcome data on PTSD symptoms, depression, anxiety, anger, and forgiveness.

DETAILED DESCRIPTION:
PTSD is a complex physiological, cognitive, emotional, and behavioral reaction to trauma comprising symptoms such as heightened arousal, emotional numbing, avoidance of trauma-related cues, and re-experiencing aspects of the trauma. Estimates indicate that 16.6% of OEF/OIF veterans returning from deployment develop PTSD (Hoge et al., 2007), much higher than the overall prevalence rate of 6.8% among adults in the United States (Kessler et al., 2005). Although efficacious treatments for PTSD are available, considerably less is known about preventing its progression from sub-threshold symptoms to full PTSD (Feldner, Manson, & Friedman, 2007). This is disconcerting because studies show that sub-threshold PTSD is a potential risk factor for the development of PTSD (e.g., Buckley, Blanchard, & Hickling, 1996; Carty, O'Donnell, & Creamer, 2006). Thus, there is a need for the development and evaluation of brief preventive interventions that can be easily and effectively implemented with individuals who have sub-threshold PTSD, defined as meeting either DSM-IV PTSD criteria B and C or B and D, but failing to meet all three, and experiencing at least one month of significant impairment (Blanchard et al., 1994).

Although treatments for PTSD such as Cognitive Processing Therapy (CPT) and Prolonged Exposure (PE) have been generally successful with individuals with full-blown PTSD (Foa et al., 1991; Monson et al., 2006; Schnurr et al., 2007), these treatments have not been systematically evaluated within a context of prevention and applied to individuals with sub-threshold symptoms. Furthermore, despite the effectiveness of available treatments for trauma symptoms, several identified barriers to treatment exist for veteran populations, particularly those who live in rural settings.

These barriers to care highlight the need for brief, cost-effective, and self-managed interventions aimed at reducing attrition, providing symptom relief, and preventing PTSD in rural and underserved populations. One potentially valuable intervention is expressive writing (i.e., writing thoughts and feelings about a significant life event). Expressive writing is associated with large improvements in psychiatric and physical symptoms and can be modified to suit the needs of specified groups (e.g., Frisina, Borod, & Lepore, 2004; Pennebaker, 2004; Smyth, 1998). Forgiving others can decrease physiological arousal (Lawler et al., 2003; Witvliet, Ludwig, & VanderLaan, 2001), depression, anxiety, and post-traumatic stress (Reed & Enright, 2006), as well as anger and substance use (Lin et al., 2004), while self-forgiveness is associated with improved quality of life and decreased mood disturbance (Friedman et al., 2007; Romero et al., 2006). Thus, a forgiveness-based writing intervention may be particularly powerful for addressing responses to trauma. Although previous studies have examined forgiveness-based writing interventions (McCullough, Root, & Cohen, 2006; Romero, 2008), none has examined the benefits of forgiveness-based writing for patients with sub-threshold PTSD symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Men and women of all racial/ethnic backgrounds between the ages of 18 and 64, seen in the identified settings (veteran participants must be OEF/OIF).
* Presence of sub-threshold PTSD as defined by Blanchard et al. (1994), related to combat experienced in the past 2 years.
* Ability to read, write, and speak English.
* Ability to attend on-site baseline and follow-up appointments.
* Ability to be contacted by phone with study reminders.

Exclusion Criteria:

* Primary psychotic disorder unrelated to PTSD.
* Impaired cognitive functioning.
* Current suicidal or homicidal intent.
* Symptoms meeting full PTSD diagnostic criteria.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-07 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
TEI-SF (Treatment Evaluation Inventory-Short Form) | One-month follow-up
CSQ-8 (Client Satisfaction Questionnaire) | One-month follow-up

SECONDARY OUTCOMES:
SCID-PTSD Module | Baseline and One-Month Follow-up
DASS-21 (Depression Anxiety and Stress Scales) | Baseline, One-week Post, and One-month Follow-up
PCL-C (PTSD Checklist- Civilian Version) | Baseline, One-week Post, and One-month Follow-up
PTCI (Posttraumatic Cognitions Inventory) | Baseline, One-week Post, One-month Follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Catherine R. Barber, PhD, Principal Investigator — MIRECC Affiliate
Locations (1):
- Michael E. DeBakey Veterans Affairs Medical Center, Houston, Texas, United States